CLINICAL TRIAL: NCT05593939
Title: Slow Age: a Randomized, Controlled Clinical Trial of Interventions to Slow Aging in Humans
Brief Title: Slow Age: Interventions to Slow Aging in Humans
Acronym: SlowAge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Elysium Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-21017723
Record Dates: First submitted 2022-09-27; First posted 2022-10-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-09

CONDITIONS: Aging
MeSH Terms: interventions — Exercise; nicotinamide-beta-riboside

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise arm (Experimental): 12 week aerobic exercise will be performed in agreement with current guidelines for exercise in older adults from the American College of Sports Medicine. A frequency of 5 days/week, totaling 150-300 min/week, performed at both moderate and vigorous intensities is chosen. This dose has a high level of evidence supporting positive effects on health- and life-span.
  Interventions: Behavioral: Exercise
- Time restricted feeding (Experimental): A 12 week fasting/feeding regiment of 16 hours fasting /8 hours feeding each day is chosen. This ratio has been shown to be tolerable in older individuals.
  Interventions: Behavioral: Time restricted feeding
- Nicotinamide riboside (Experimental): Previous clinical trials have shown that an nicotinamide riboside dose up to 2 g/day is well tolerated with no treatment-emergent adverse events reported so far and with efficacy on our primary outcome measurement. A dose of 2 g/day NR is therefore chosen and will be split in two: 1 g in the morning and 1 g in the evening.
  Interventions: Dietary Supplement: Nicotinamide riboside
- Control (No Intervention): A control group with no intervention.

INTERVENTIONS:
Behavioral: Exercise — Participants randomized to the EXE group will perform aerobic exercise five days per week, totaling 150-300 min/week, at moderate to vigorous intensities i.e., ~60-90% heart rate (HR) max. Participants randomized to the EXE group will perform aerobic exercise five days per week, totaling 150-300 min/week, at moderate to vigorous intensities i.e., ~60-90% heart rate (HR) max. Exercise intensity and duration will gradually increase up until week 3 to habituate the participants to the exercise. The training modality will change to reduce the risk of injuries and may be impacted by individual preferences to increase adherence. The training can be performed individually or in groups of 4-6 participants, depending on the geographical locations of the participants home address, and on the current recruitment rate.
  Arms: Exercise arm
Behavioral: Time restricted feeding — Participants randomized to the time restricted feeding group will be instructed to abstain from any caloric intake during the targeted fasting window of 16 continuous hours and consume ad libitum during the eating window of 8 hours.
  Arms: Time restricted feeding
Dietary Supplement: Nicotinamide riboside — Participants randomized to the NR group will be instructed to take the administered tablets once in the morning (1 g) and once in the evening (1 g), in both cases with a meal.
  Arms: Nicotinamide riboside

SUMMARY:
The proportion of older individuals is growing, and it is therefore important to investigate ways to promote healthy aging. Exercise is one of the most studied interventions and is known to have a variety of health benefits. Dietary interventions have also shown encouraging results, with intermittent fasting being a promising anti-aging intervention. Likewise, dietary supplementation with precursors that can increase the central metabolite nicotinamide dinucleotide (NAD+) has powerful effects on aging at least in model organisms. Although physical exercise is known to increase health-span, the effects of these latter dietary interventions on aging lacks evidence in humans.

This is a randomized, controlled trial of interventions to slow aging in humans. Healthy older individuals will be randomized into either an aerobic exercise (EXE), time-restricted feeding (TRF), nicotinamide riboside (NR), or control group and followed for twelve weeks. Changes in biomarkers of aging will be assessed before and after the intervention. It is hypothesized that the interventions provide similar, superior benefits to these markers when compared to placebo.

Primary Outcome: Interleukin-6 levels. Secondary Outcomes: CRP, TNF-α, NAD+, hematologic age, epigenetic age (DNA methylation), transcriptomic age (RNA-sequencing), functional age (handgrip strength, gait speed), body composition, vocal age, and photo age

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Aged ≥ 65 years
4. In good general health

Exclusion Criteria:

1. Inability or unwillingness to take oral supplements
2. Inability or unwillingness to adhere to the fasting regiment
3. Inability or unwillingness to perform the prescribed physical exercise
4. Current smoker or use of any nicotine products within 10 years
5. Chronic use of supplements containing vitamin B or nicotinamide riboside
6. Treatment with another investigational drug or other intervention within 1 year
7. Cancer diagnosis within last 5 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 levels in plasma | Day 1 compared to day 84

SECONDARY OUTCOMES:
Concentration of CRP in plasma | Day 1 compared to day 84
Concentration of TNF-α in plasma | Day 1 compared to day 84
Concentration of NAD in whole blood | Day 1 compared to day 84
Change in fat mass | Day 1 compared to day 84
  Measured using bio-impedance
Change in lean mass | Day 1 compared to day 84
  Measured using bio-impedance
Grip strength | Day 1 compared to day 84
Gait speed | Day 1 compared to day 84
  Measured over 4 meters.
Predicted age (DNA methylation) | Day 1 compared to day 84
  From PBMCs
Predicted age (Blood age) | Day 1 compared to day 84
  From 33 blood parameters
Predicted age (Transcriptomics) | Day 1 compared to day 84
  From RNA seq of PBMCs
Predicted age (voice) | Day 1 compared to day 84
  From voice recordings
Predicted age (photo) | Day 1 compared to day 84
  From a portrait photo

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
This is not possible under current data protection rules.